CLINICAL TRIAL: NCT06965426
Title: Effect of Lutein, Zeaxanthin, and Meso-Zeaxanthin Supplementation on Skin Carotenoid Concentration: A Six-Month, Placebo-Controlled Crossover Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insight Eyecare Specialties, Inc. dba Vision Source Eyecare, (Other)
Collaborators: MacuHealth (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: VSE001
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Macular Degenerative Disease
Keywords: Carotenoids; Macular degeneration; MacuHealth
MeSH Terms: conditions — Macular Degeneration | interventions — Lutein; Zeaxanthins

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Placebo vs. Vitamin will be masked to patient and investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MacuHealth Supplementation (Active Comparator): Lutein, Zeaxanthin, and Meso-Zeaxanthin Supplementation
  Interventions: Other: Lutein, Zeaxanthin, and Meso-Zeaxanthin Supplementation
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Lutein, Zeaxanthin, and Meso-Zeaxanthin Supplementation

INTERVENTIONS:
Other: Lutein, Zeaxanthin, and Meso-Zeaxanthin Supplementation — Lutein, Zeaxanthin, and Meso-Zeaxanthin Supplementation
  Other Names: MacuHealth

SUMMARY:
To compare skin carotenoid scores over 12 weeks of individuals randomized to placebo or MacuHealth and comparing that to a 12 week crossover evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-50 years old of any sex and any race.
* Willing to comply with the protocol instructions.
* Has read (or has had read to), understood, and signed an Informed Consent.

Exclusion Criteria:

* Current Smoker
* Pregnant, plan to become pregnant or breastfeeding
* History of any non-controlled disease states including diabetes, cancer, heart diseases ETC (we need to confirm this with previous protocols) BMI greater than 30
* Currently taking MacuHealth or similar supplements or previous use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Carotenoid concentration | 6 months
  Change in skin carotenoid concentration over supplementation vs. placebo exposure durations.

CONTACTS AND LOCATIONS:
Locations (1):
- Vision Source, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided